CLINICAL TRIAL: NCT04631835
Title: A Phase 1, Open-label, Multicenter Study to Evaluate Safety, Tolerability, Pharmacokinetics, and Efficacy of Single and Multiple Doses of Oral Administration of HS-10352 in Patients With Locally Advanced or Metastatic Breast Cancer Progressing After Standard Therapy
Brief Title: Phase I Study of the HS-10352 in Patients With Advanced Breast Cancer
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jiangsu Hansoh Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HS-10352-101
Record Dates: First submitted 2020-11-09; First posted 2020-11-17 (Actual); Last update posted 2022-06-15 (Actual); Status verified 2022-06

CONDITIONS: Breast Cancer
Keywords: dose-escalation; advanced solid tumors; estrogen receptor positive breast cancer; PIK3CA gene mutation
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HS-10352 (Experimental): There are five escalating dose cohorts
  Interventions: Drug: HS-10352

INTERVENTIONS:
Drug: HS-10352 — Participants will receive single dose of HS-10352 on Day 1 of Cycle 1 followed by once daily from Day 8 of Cycle 1. (Cycle length: 35 days for Cycle 1 and 28 days for all other cycles). Participants will continue treatment until the end of the study in the absence of unacceptable toxicities and unequivocal disease progression.

SUMMARY:
HS-10352 is a highly potent and selective small molecule inhibitor of phosphoinositide 3-kinase (p110α). In preclinical studies, it demonstrated strong activity against PI3K p110α in vitro and in vivo, and inhibited tumor cell growth. The first-in-human trial is conducted to assess the maximum tolerated dose (MTD) and dose limiting toxicity (DLT), to evaluate the pharmacokinetics, safety and preliminary anti-tumor activity of HS-10352 at single dose and multiple doses.

DETAILED DESCRIPTION:
This is a phase I, open-label, multicenter study to evaluate safety, tolerability, pharmacokinetics, and efficacy of single and multiple doses of oral administration of HS-10352 in patients with locally advanced or metastatic breast cancer with hormone receptor (HR) positive and epidermal growth factor receptor 2 (HER2) negative who have progressed following prior therapy. There is a dose-escalation study, which is designed to evaluate the safety, tolerability, and pharmacokinetics of single dose and multiple doses of HS-10352 given once every day (QD). An alternative dosing schedule of twice every day (BID) may be investigated if the drug clearance of HS-10352 is faster than anticipated.

All patients will be carefully followed for adverse events during the study treatment and for 28 days after the last dose of study drug. Subjects of this study will be permitted to continue therapy with assessments for progression once every 8 weeks, if the product is well tolerated and the subject has stable disease or better. As the disease progresses, survival follow-up is recommended bimonthly.

ELIGIBILITY:
Inclusion Criteria:

1. Men or women aged more than or equal to (≥) 18 years, and less than (<) 75 years.
2. HR+ HER2- locally advanced or metastatic breast cancer patients confirmed by histology or cytology for who that standard treatment is invalid, unavailable or intolerable.
3. Patients have at least one target lesion according to RECEST 1.1. The requirements for target lesions are: measurable lesions without local treatment such as irradiation, or with definite progress after local treatment, with the longest diameter ≥ 10 mm in the baseline period (in case of lymph nodes, the shortest axis ≥ 15 mm is required)
4. ECOG performance status was 0-1 and did not deteriorate in the previous 2 weeks.
5. Estimated life expectancy greater than (>) three months.
6. Females should be using adequate contraceptive measures throughout the study; should not be breastfeeding at the time of screening, during the study and until 3 months after completion of the study; and must have evidence of non-childbearing potential.
7. Sign Informed Consent Form.

Exclusion Criteria:

1. Treatment with any of the following:

   1. Previous or current treatment with PI3K, AKT or mTOR inhibitors.
   2. Any cytotoxic chemotherapy, investigational agents within 21 days of the first dose of study drug; anticancer drugs which have been received within 14 days before the first administration.
   3. Radiotherapy with a limited field of radiation for palliation within 2 weeks of the first dose of study drug, or patients received more than 30% of the bone marrow irradiation, or large-scale radiotherapy within 4 weeks of the first dose.
   4. Major surgery (including craniotomy, thoracotomy, or laparotomy, etc.) within 4 weeks of the first dose of study drug.
2. Inadequate bone marrow reserve or organ function.
3. Uncontrolled pleural effusion or ascites or pericardial effusion.
4. Known and untreated, or active central nervous system metastases.
5. History of primary or secondary diabetes.
6. History of acute or chronic pancreatitis
7. Refractory nausea, vomiting, or chronic gastrointestinal diseases, or inability to swallow the study drug that would preclude adequate absorption of HS-10352.
8. History of hypersensitivity to any active or inactive ingredient of HS-10352 or to drugs with a similar chemical structure or class to HS-10352.
9. Judgment by the investigator that the patient should not participate in the study if the patient is unlikely to comply with study procedures, restrictions, and requirements.
10. Any disease or condition that, in the opinion of the investigator, would compromise the safety of the patient or interfere with study assessments.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2020-09-08 (Actual); Primary Completion 2023-04-30 (Estimated); Study Completion 2023-08-31 (Estimated)

PRIMARY OUTCOMES:
Number of subjects with any dose limiting toxicity (DLT) | From the single dose to the last dose of the first cycle defined as 28 days of multiple dosing (35 days).
  DLT is defined as one of the following HS-10352 related adverse event (AE) that occurs during the DLT period, excluding AE assessed by investigator exclusively related to subject's underlying disease or medical condition (graded according to the NCI Common Terminology Criteria for Adverse Events (CTCAE), Version 5.0):
To determine the maximum tolerated dose (MTD) | From the single dose to the last dose of the first cycle defined as 28 days of multiple dosing (35 days).
  MTD was defined as the previous dose level at which 2 of 2 subjects or 2 out of 6 subjects experienced a DLT.

SECONDARY OUTCOMES:
Incidence and severity of treatment-emergent adverse events | From baseline until 28 days after the last dose
  Assessed by number and severity of adverse events as recorded on the case report form, vital signs, laboratory variables, physical examination, electrocardiogram, RECIST1.1, and NCI CTCAE v5.0.
Observed maximum plasma concentration (Cmax) after single dose of HS-10352 | From pre-dose to 120 hours after single dose on Day 1
  In the study of single-dose, Cmax will be obtained following administration of a single oral dose of HS-10352 on Day 1 to Day 6.
Observed maximum plasma concentration (Cmax ss) after multiple dose of HS-10352 | From pre-dose to 24 hours after the first dose of multiple dosing on Day 1 of the second 28-Day cycle of therapy
  At multiple-dose, Cmax ss will be obtained on Day 1 of dosing in the second 28-Day cycle of therapy.
Time to reach maximum plasma concentration (Tmax) after single dose of HS-10352 | From pre-dose to 120 hours after single dose on Day 1
  In the study of single-dose, Tmax will be obtained following administration of a single oral dose of HS-10352 on Day 1 to Day 6.
Time to reach maximum plasma concentration (Tmax) after multiple dose of HS-10352 | From pre-dose to 24 hours after the first dose of multiple dosing on Day 1 of the second 28-Day cycle of therapy
  At multiple-dose, Tmax will be obtained on Day 1 of dosing in the second 28-Day cycle of therapy.
Apparent terminal half-life (t1/2) after single dose of HS-10352 | From pre-dose to 120 hours after single dose on Day 1
  Apparent terminal half-life is the time measured for the concentration to decrease by one half. Terminal half-life calculated by natural log 2 divided by λz.
Area under plasma concentration versus time curve from zero to the 24-hour sampling time (AUC0-24) after single dose of HS-10352 | From pre-dose to 24 hours after single dose on Day 1
  Area under the plasma concentration versus time curve from time zero to the 24-hour sampling time at which the concentration was at or above the lower limit of quantification (LLQ). AUC0-24 was to be calculated according to the mixed log-linear trapezoidal rule.
Area under plasma concentration versus time curve from zero to last sampling time (AUC0-t) after single dose of HS-10352 | From pre-dose to 120 hours after single dose on Day 1
  Area under the plasma concentration versus time curve from time zero to the last sampling time t at which the concentration was at or above the lower limit of quantification (LLQ). AUC0-t was to be calculated according to the mixed log-linear trapezoidal rule.
Area under the plasma concentration versus time curve from time zero to infinity (AUC0-∞) after single dose of HS-10352 | From pre-dose to 120 hours after single dose on Day 1
  AUC0-∞ was calculated by combining AUC0-t and AUCextra. AUCextra represents an extrapolated value obtained by Clast/ λz, where Clast is the calculated plasma concentration at the last sampling time point at which the measured plasma concentration is at or above the LLQ and λz is the apparent terminal rate constant determined by log-linear regression analysis of the measured plasma concentrations of the terminal log-linear phase.
To further evaluation of the anti-tumor activity of HS-10352 by assessment of objective response rate (ORR) | From the date of first occurrence of complete response (CR) or partial response (PR) on 2 consecutive occasions (≥4 weeks), until the date of disease progression or withdrawal from study, approximately 3 years
  Anti-tumor efficacy will be assessed by best radiographic response based on Response Evaluation Criteria in Solid Tumors at baseline (Day -28 to -1). For patients that continue on repeating 28-Day cycles after the primary evaluation period, progression will be assessed after each 8 weeks of therapy. ORR is defined as the percentage of patients with a complete response (CR) or partial response (PR) that was confirmed at a subsequent scan at least 4 weeks later, as assessed according to RECIST version 1.1.
Disease control rate of HS-10352 | From the first occurrence of confirmed CR or PR or SD until the date of disease progression or withdrawal from study, approximately 3 years
  Objective response was assessed by RECIST 1.1 thereby to evaluate disease control rate. Disease control was deﬁned as the percentage of patients who have a best overall response (confirmed CR, PR, or stable disease for at least 6 weeks).
Deepness of response of HS-10352 | From the date of enrollment until the date of disease progression or death, approximately 3 years
  Objective response was assessed by RECIST 1.1 thereby to evaluate deepness of response. Depth of response was defined as the relative change in the sum of the longest diameters of RECIST target lesions at the nadir in the absence of new lesions, or progression of non-target lesions compared with baseline.
Progression-free survival of HS-10352 | From the date of enrollment until the date of disease progression or death from any cause, approximately 3 years
  Progression of tumor was assessed by RECIST 1.1 thereby to evaluate progression free survival. Progression-free survival was deﬁned as the time from date of ﬁrst dose until the documentation of objective disease progression (PD) or death from any cause in the absence of progression (whichever occurred first), regardless of whether they subsequently received non-study anti-cancer therapy.
Overall survival of HS-10352 | From the date of enrollment until the date of death from any cause, approximately 5 years
  Overall survival was deﬁned as the time from date of ﬁrst dose until the documentation of death from any cause.

CONTACTS AND LOCATIONS:
Locations (3):
- China (3):
  - SUN YAT-SEN Memorial Hospital, Guanzhou, Guangdong
  - Hunan Cancer Hospital, Changsha, Hunan
  - Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality

REFERENCES:
- [Derived] Ouyang Q, Wang Y, Zhang J, Wu Q, Wei H, Li C, Qian X, Hu X. HS-10352 in hormone receptor-positive, HER2-negative advanced breast cancer: A phase 1 dose-escalation trial. Cancer Med. 2023 Dec;12(24):21849-21860. doi: 10.1002/cam4.6755. Epub 2023 Dec 1. PMID 38037839